CLINICAL TRIAL: NCT05023460
Title: Treatment of Chronic Cluster Headache (Horton's Headache) with Transcutaneous Electrical Nerve Stimulation and Occipital Nerve Stimulation
Brief Title: Treatment of Chronic Cluster Headache with TENS and ONS
Acronym: HortONS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Danish Headache Center (Other)
Responsible Party: Principal Investigator, Ida Stisen Fogh-Andersen, PhD fellow, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HortONS
Record Dates: First submitted 2021-07-27; First posted 2021-08-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Chronic Cluster Headache; Primary Headache Disorder; Headache; Cluster Headache; Pain; Cephalgia; Trigeminal Autonomic Cephalgia
Keywords: Occipital nerve stimulation; Neuromodulation; Transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Cluster Headache; Headache Disorders, Primary; Headache; Pain; Trigeminal Autonomic Cephalalgias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Paresthesia-free (burst) ONS (Active Comparator): Implanted lead and impulse generator (IPG), paresthesia-free (burst) active stimulation.
  Lead implanted subcutaneously over greater occipital nerves. Implanted IPG capable of providing paresthesia-free stimulation continuously.
  Interventions: Device: Paresthesia-free (burst) ONS
- Placebo (Placebo Comparator): Implanted lead and IPG, deactivated.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Paresthesia-free (burst) ONS — Stimulation intensity target of 60% of paresthesia threshold.
  Arms: Paresthesia-free (burst) ONS
Device: Placebo — ONS system deactivated
  Arms: Placebo

SUMMARY:
The study is an investigator-initiated, prospective, randomized, placebo-controlled, double blind clinical trial that aims to investigate the effect of transcutaneous electrical nerve stimulation (TENS) and occipital nerve stimulation (ONS) on attack frequency and severity in patients with chronic cluster headache (CH).

Study outline

Month 1: Baseline. Establishment of a baseline profile of the participants CH attacks (severity, duration, medicine utilization etc), health-related quality of life (QoL) and symptoms of anxiety and depression. No active treatment. Follow-up visit after 30 days.

Months 2-4: TENS period. All participants will receive TENS-treatment. Clinical follow-up visit by the end of month four.

Months 5-7: Double-blinded, randomized experimental period. All participants will have an ONS-system (lead, impulse generator) implanted and will be randomized 1:1 to receive either 1) burst (paresthesia-free) ONS or 2) placebo (deactivated ONS system). Clinical follow-up visit by the end of month seven.

Months 8-10: Open label period. All participants will receive tonic (conventional, paresthesia-inducing) ONS.

Clinical follow-up visit by the end of month ten.

During every study phase each participant will fill out a weekly electronic headache registration as well as answering questionnaires regarding health-related quality of life and symptoms of anxiety and depression before every follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Signed informed written consent
3. Diagnosed with chronic CH according to the ICHD-3 criteria
4. 15 or more CH attacks per month
5. Stable use of preventive headache medication one month prior to enrollment

Exclusion Criteria:

1. Other ongoing neuromodulation therapy
2. Current alcohol and/or drug abuse
3. Severe psychiatric disorder
4. Other chronic primary or chronic secondary headache disorder (e.g. chronic migraine)
5. Major posterior neck surgery in C2-C3 level and above
6. Pregnancy
7. Treatment with oral steroids or GON injection within one month of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
30% reduction in CH attack frequency with TENS- and ONS-treatment | Primary evaluation through month 4 (TENS) and 7 (ONS, blinded)
  Proportion of participants with a positive treatment outcome of a 30% reduction in CH attack frequency compared to baseline.
  A CH attack is here defined as any attack recognised by the patient as a CH attack.
Incidence of treatment-emerged adverse events [safety] in TENS treatment | Evaluation at month 4
  Treatment related adverse events and adverse device effects will be registered on an ongoing basis. Serious events will be handled immediately.
Incidence of treatment-emerged adverse events [safety] in ONS treatment | Evaluation at month 7 (burst ONS) and 10 (tonic ONS)
  Treatment related adverse events and adverse device effects will be registered on an ongoing basis. Serious events will be handled immediately.

SECONDARY OUTCOMES:
30% reduction of pain intensity in CH attacks | Through month 4, 7 and 10
  Weekly self reported pain intensity on a numeric rating scale from 0-10 with 0 being "no pain" and 10 "the worst possible pain".
  Proportion of participants with a positive treatment outcome of a 30% reduction in pain intensity during CH attacks compared to baseline.
Feasibility of TENS as a predictor for the efficacy of ONS treatment | Through month 4 and 10
  Comparison will be made of headache data from the last month of treatment with TENS and tonic ONS, respectively, to evaluate whether a 30% reduction in CH attack duration with TENS-treatment correlates to a 30% reduction in CH attack duration with ONS-treatment.
Non-inferiority study: Burst ONS versus tonic ONS | Through month 7 and 10
  Comparing treatment outcome of burst ONS and tonic ONS.
Patient-perceived Global Impression of Change (PGIC) | At month 4, 7 and 10
  The number of participants who rates their condition 'much improved' or 'very much improved' as assessed by PGIC.
Reduction in background headache | At month 4, 7 and 10
  Proportion of participants reporting a reduction in background headache. A positive treatment outcome will be defined as a two-point improvement on a four-point scale compared to baseline.
Hospital anxiety and depression scale (HADS) | At month 4, 7 and 10
  HADS is a self-assessment questionnaire consisting of seven items each for depression and anxiety sub-scales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level.
  HADS score will be evaluated at every follow up and compared to baseline.
Health-related quality of life (EuroQoL 5D-5L) | At month 4, 7 and 10
  The EQ 5D-5L is a well-established measure of health-related quality of life that is quantified as a utility (a measure of quality of life between 0 and 1) based on a danish value set. Furthermore a total score that ranges from 0-100 (visual analog scale), a higher score indicates better health-related quality of life.
Self reported sleep quality | At month 4, 7 and 10
  Proportion af participants reporting a positive treatment outcome defined as a two-point improvement on a four-point scale compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ida S Fogh-Andersen, MD PhD fellow, Principal Investigator — University of Aarhus; Kaare Meier, MD PhD, Study Director — University of Aarhus; Jens Christian H Sørensen, MD PhD DMSc, Study Chair — University of Aarhus; Rigmor H Jensen, MD PhD DMSc, Study Chair — Danish Headache Centre
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fogh-Andersen IS, Petersen AS, Jensen RH, Sorensen JCH, Meier K. Transcutaneous electrical nerve stimulation of the occipital nerves as treatment for chronic cluster headache. Headache. 2025 Jun;65(6):973-982. doi: 10.1111/head.14889. Epub 2024 Dec 20. PMID 39703191
- [Derived] Fogh-Andersen IS, Sorensen JCH, Petersen AS, Jensen RH, Meier K. The HortONS study. Treatment of chronic cluster headache with transcutaneous electrical nerve stimulation and occipital nerve stimulation: study protocol for a prospective, investigator-initiated, double-blinded, randomized, placebo-controlled trial. BMC Neurol. 2023 Oct 21;23(1):379. doi: 10.1186/s12883-023-03435-9. PMID 37865755